CLINICAL TRIAL: NCT01688024
Title: Phase 2 Study of Mitomycin C Therapy for Biliary Strictures in Patients With Primary Sclerosing Cholangitis
Brief Title: Mitomycin C Therapy for Patients With Primary Sclerosing Cholangitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li, Zhiping, M.D. (Individual)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00052685
Record Dates: First submitted 2012-09-10; First posted 2012-09-19 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: mitomycin C
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Mitomycin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin C (Experimental): Up to 10 mg administered during each standard of care endoscopic retrograde cholangiography. No more than five mitomycin C applications per every twelve months will be given.
  Interventions: Drug: Mitomycin C
- Normal saline (Placebo Comparator): Given during each standard of care endoscopic retrograde cholangiography. No more than five normal saline applications per every twelve months will be performed.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Mitomycin C
  Arms: Mitomycin C
Drug: Normal saline
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of mitomycin C in the treatment of primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Previously established diagnosis of primary sclerosing cholangitis

Exclusion Criteria:

* American Society of Anesthesiologists class 4 or greater
* Serum creatinine >= 1.7 mg/dL, eGFR <= 30 mL/min, or dialysis dependence
* Serum hemoglobin <= 7 g
* Left ventricular ejection fraction <= 30%
* Dyspnea with minimal exertion (or supplemental oxygen dependence)
* History of bone marrow disease
* Prior recipient of organ transplantation
* Ongoing chemotherapy
* Obstruction of the upper GI tract
* Pregnant or lactating
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Effect on Disease Prognosis as Determined by the Mayo Natural History Model for Primary Sclerosing Cholangitis | Two years

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | Two years
Frequency of Endoscopic Interventions Needed to Manage Disease-related Complications | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Zhiping Li, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States